CLINICAL TRIAL: NCT05123105
Title: Effect of Dry Cupping and Ischemic Compression on the Trigger Point on the Upper Trapezius Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Agnieszka Zdrodowska, academic researcher, doctor of science, Józef Piłsudski University of Physical Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SKE 01-03/2021
Record Dates: First submitted 2021-10-23; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: ischemic compression; cupping; algometer; trapezius muscle
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Cupping Therapy; Acupressure

STUDY DESIGN:
Intervention Model Description: Each person participated in three tests with an interval of approximately one week between them. The following study protocol was followed; (short version)
  1. cupping therapy;
     - a minimum interval of 7 days;
  2. control test;
     - a minimum interval 7 days;
  3. ischemic compression.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Each person participated in three tests with an interval of approximately one week between them.
  Interventions: Other: 1) cupping therapy; Other: 2) control test (no intervention); Other: 3) ischemic compression

INTERVENTIONS:
Other: 1) cupping therapy — The participant lay on his front on a couch. The examiner applied a plastic cup on a pre-marked trigger point, suctioned it with a mechanical pump and left it for 2 minutes. This was a stationary application with medium suction force. Therapy was performed on both sides. Measurements were taken before and 2 minutes after the therapy.
Other: 2) control test (no intervention) — The participant lay on his front on a couch for 4 minutes without any activity and without anyy intervention. Measurements were taken before and after the session.
Other: 3) ischemic compression — The participant lay on his front on a couch. The researcher applied pressure to a pre-marked trigger point using the thumb for 2 minutes until tissue resistance was felt. This included 60-second compression and after a break of a few seconds, another 60 seconds of compression. Therapies were performed on each side. Measurements were taken before and 2 minutes after the therapy.

SUMMARY:
Ischemic compression is considered the fastest and most common method for providing relief in trigger point therapy, whereas cupping therapy is not a method often used for this purpose. The muscle that has a great impact on tension-type headaches and neck pain is the trapezius, whose upper fibres are where the most common trigger point in the back is located.

The aim of this study was to evaluate and compare the effectiveness of single ischemic compression and single dry cupping therapy on the most common trigger point, on the descending part of the trapezius muscle.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* student of The Józef Piłsudski University of Physical Education in Warsaw
* written consent to participate in the study

Exclusion Criteria:

* past or current injury to the trapezius.
* past or current injury of the cervical spine limiting mobility of this segment.
* broken skin at the examination site.
* cardiological disease and use of blood pressure medication, histamine medication and analgesics
* elevated body temperature, illness symptoms and a period of convalescence.
* a missed anti-Covid procedure before each examination.
* inability to find trigger points.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-23 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold test (PPT) | changes from baseline in pain pressure threshold at 2 minutes after the session
  The trigger points of the upper section of the trapezius on the right and left sides were determined by palpation and were also indicated using a marker. A Wagner FDX 50 Force Gage algometer was applied to the trigger point. The pressure force was increased by 1kg/cm2/s until the patient felt pain, which was the pain pressure threshold (PPT) measured in kg/cm2. The test was performed on both sides. The test was performed twice on each side - before and 2 minutes after the session.
Cervical spine mobility test | changes from baseline in cervical spine mobility at 2 minutes after the session
  Each examination began in a sitting position with a cervical spine mobility test. The following bone points were marked on the participants' skin using a marker: spinous process of the 7th cervical vertebra, external occipital protuberance, the top of the chin, the jugular notch of the sternum, the mastoid of the temporal bone, and the acromion process of the scapula. Next, a linear measurement of the range of motion was performed using a tape measure to ascertain the distance between the marked points in the initial position and after the active movement for flexion (forward bending), extension (backward bending), lateral bending and rotation to both sides, respectively. The mobility was determined by the difference of the two measurements. The test for each movement (i.e. flexion (forward flexion), extension (backward flexion), lateral flexion and both sides rotation) was performed twice - before and 2 minutes after the session.

SECONDARY OUTCOMES:
Height | Measurements were taken before the first session
  Height measured in meters
Weight | Measurements were taken before the first session
  Weight measured in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Zdrodowska, PH.D, Principal Investigator — Józef Piłsudski University of Physical Education in Warsaw
Locations (1):
- Józef Piłsudski University of Physical Education in Warsaw, Warsaw, Masovian Voivodeship, Poland